CLINICAL TRIAL: NCT01560702
Title: Endoscopic Injection of Autologous Blood Versus Diluted Epinephrine for Control of Actively Bleeding Gastroduodenal Ulcers
Brief Title: Comparative Study of Autologous Blood Injection Versus Diluted Epinephrine in Treating Actively Bleeding Gastroduodenal Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Moahmed Hassan Emara, Lecturer, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#:278/12-3-2012
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Blood, Injection, Injury Type Phobia; Gastrointestinal Ulcer Haemorrhage; Adverse Reaction to Epinephrine
Keywords: autologous blood; epinephrine; endoscopy; ulcer; hemostasis
MeSH Terms: conditions — Ulcer | interventions — Epinephrine; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous blood (Active Comparator): Patients will be injected by autologous blood at the edge of actively bleeding ulcer
  Interventions: Biological: Blood
- Epinephrine injection (Other): Patients will be injected by diluted epinephrine at the edge of actively bleeding ulcer
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: Epinephrine — 10-30 cc of 1/10000 diluted epinephrine will be injected at edges of an actively bleeding ulcer.
  Arms: Epinephrine injection
Biological: Blood — 5-20 cc autologous blood immediately withdrawn from the patient will be injected at edges of the actively bleeding ulcer.
  Arms: Autologous blood

SUMMARY:
Endoscopic injection of autologous blood can control bleeding from gastroduodenal ulcers.

DETAILED DESCRIPTION:
To test the hypothesis that endoscopic injection of autologous blood is superior to endoscopic injection of diluted epinephrine in controlling bleeding from gastroduodenal ulcers.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients with gastroduodenal ulcer

Exclusion Criteria:

* Patients with non ulcer bleeding.
* Patients with malignancy.
* Patients with bleeding disorders or under coagulation therapy.
* Patients with known allergy to epinephrine.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
hemostasis from the ulcer after injection and/or stoppage of haematemesis and melena one day after the procedure. | 12 months

SECONDARY OUTCOMES:
development of re-bleeding after 24 hours after the procedure (occurrence of hematemesis or melena or drop of hemoglobin level >2gm/dl). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Emara, MD, Principal Investigator — Tropical Medicine Department, Faculty of Medicine, Zagazig University, Zagazig, 44519, Egypt
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqia Province, Egypt

REFERENCES:
- See also: Our Department official journal — http://mis.zu.edu.eg/ajied/home.aspx
- See also: Our Hospital — http://www.hosp.zu.edu.eg/